CLINICAL TRIAL: NCT07188961
Title: The Effect of Kinesiologic Taping on Trunk Control and Balance in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Ozden Baskan, Assistant Professor, Istanbul Rumeli University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-53938333-050-45047
Record Dates: First submitted 2025-08-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy (CP); Balance; Kinesiology Taping; Spasticity
Keywords: cerebral palsy; balance; trunk
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gruop 1 (Experimental): Kinesiologic taping was performed a total of four times, once a week.
  Interventions: Other: kinesiologic taping

INTERVENTIONS:
Other: kinesiologic taping — This intervention is distinguished from other studies by its combined assessment of trunk and extremity kinesiology taping in children with both hemiplegic and diplegic cerebral palsy over a four-week period.

SUMMARY:
Title: Effects of Kinesiology Taping on Motor Function, Balance, and Spasticity in Children with Hemiplegic and Diplegic Cerebral Palsy: A Four-Week Study Study Type: Interventional (Clinical Trial) Study Design: Single-group, pre-post design Condition: Cerebral Palsy (Hemiplegic and Diplegic) Intervention: Kinesiology taping applied to trunk and extremity muscles over four weeks

Primary Outcome Measures:

Trunk and joint range of motion (ROM) Manual muscle testing (MMT) of the trunk Spasticity assessment using the Modified Ashworth Scale (MAS)

Secondary Outcome Measures:

Gross Motor Function Classification System (GMFCS) Functional Independence Measure for children (WeeFIM) Paediatric Berg Balance Scale (PBS) Sitting Assessment Scale (SAS) Study Duration: 4 weeks Sample Size: 30 children (aged X-Y years) with hemiplegic or diplegic cerebral palsy Pre- and post-intervention assessments were conducted. The study evaluates the short-term effects of kinesiology taping on motor function, spasticity, balance, and trunk control.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with diparetic or hemiparetic cerebral palsy by a specialist physician;
* Regular participation in physiotherapy sessions
* Gross Motor Function Classification System (GMFCS) level 1, 2, or 3; Age between 2 and 18 years

Exclusion Criteria:

* Children who have not attended physiotherapy sessions in the past six months,
* Use of a trunk brace,
* GMFCS level 4 or 5,
* History of allergic reaction to kinesiology tape,
* History of surgery within the past three months

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure for children (WeeFIM) | The study continued for 5 months. But we assessed Children in 0. week and 4. week.
  There are a total of 18 questions. Scoring ranges from 1 to 7.a high score indicates increased independence
Paediatric Berg Balance Scale (PBS) | The study continued for 5 months. But we assessed Children in 0. week and 4. week.
  This scale consists of 14 sections. Each section is scored from 0 to 4. A high score indicates increased balance.
Sitting Assessment Scale (SAS) | The study continued for 5 months. But we assessed Children in 0. week and 4. week.
  It uses a scale of 1 (none), 2 (poor), 3 (moderate), and 4 (good) for children with cerebral palsy (CP). A high score indicates increased sitting balance.

SECONDARY OUTCOMES:
Spastisity | The study continued for 5 months. But we assessed Children in 0. week and 4. week.
  Spastisity was evaluated with Modified Ashworth Scale. Each section is scored from 0 to 4. A high score indicates hih spasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ozden Baskan, Istanbul, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT07188961/Prot_000.pdf